CLINICAL TRIAL: NCT06656273
Title: Science-based Habit Formation App As an Adjunct to the National Diabetes Prevention Program (DPP) Lifestyle Change Program (LCP) to Increase Engagement, Participation and Outcomes of Underserved Populations and Others Eligible for the DPP LCP
Brief Title: Habit Building Software Application to Increase Engagement of Vulnerable Populations in the National Diabetes Prevention Program (NDPP) Lifestyle Change Program (LCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute for Iterative Thinking (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1300367-20210112; 75D30119C06604 (Other Grant/Funding Number: The Centers for Disease Control and Prevention)
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FT LCP (Experimental)
  Interventions: Behavioral: FT LCP
- Standard LCP (No Intervention)

INTERVENTIONS:
Behavioral: FT LCP — FT LCP is a behavior change software application, used as an adjunct to the standard National Diabetes Prevention Program
  Arms: FT LCP

SUMMARY:
The goal of this clinical trial is to learn whether a companion software application can improve program engagement in the National Diabetes Prevention Program in adults with prediabetes. The main question[s] it aims to answer [is/are]:

Do participants using the software application (the intervention group) have better engagement with the Diabetes Prevention Program than those who do not use the companion software application (the control group)? Are participants using the software application (the intervention group) more likely to stay in the Diabetes Prevention Program longer than those who do not use the companion software application (the control group)?

Participants are those who have signed up for their local Diabetes Prevention Program and agree to be in the study.

ELIGIBILITY:
Inclusion Criteria:

* is eligible for and enrolls in a live or distance LCP at a designated study site during the enrollment period of the study
* has a smartphone or other device able to engage with the FT LCP app
* can read basic 5th grade English, as used in the FT LCP app

Exclusion Criteria:

* Cohorts and sites enrolled in concurrent, similar health app-based studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Engagement | From enrollment to end of the Lifestyle Change Program, up to 12 months.
  The primary measure for participant engagement will be the number of classes attended by a participant.
Retention | From enrollment to end of the Lifestyle Change Program, up to 12 months.
  The primary measure for retention will be the percentage of participants that remain enrolled in the LCP at the end of the study period.
Efficacy | From enrollment to end of the Lifestyle Change Program, up to 12 months.
  The primary measure of efficacy will be the percentage of participants who reach the LCP goal of ≥5% weight loss by the end of the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Institute of Iterative Thinking, Felton, California, United States

IPD SHARING:
Plan to Share IPD: No